CLINICAL TRIAL: NCT04031612
Title: Prospective and Retrospective Neoadjuvant Breast Cancer Database
Brief Title: Neoadjuvant Database
Acronym: NEOADJ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: AB2009SEIN
Record Dates: First submitted 2019-07-01; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Neoadjuvant Treatment in Breast Cancer
Keywords: Cancer; Breast, Neoadjuvant
MeSH Terms: conditions — Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant Breast Cancer: Patients undergoing neoadjuvant therapy for breast cancer
  Interventions: Drug: Neoadjuvant therapy

INTERVENTIONS:
Drug: Neoadjuvant therapy — Neoadjuvant therapy

SUMMARY:
The NEOADJ Database base contains data collected during the regular clinical patient management (sociodemographic, clinical, pathological, radiological, biological, disease evolution...). This database allows easy access to information in a centralized and structured way.

This cohort is used to gather insights for research purposes. All data collected come from medical files of patients managed at Centre Georges Francois Leclerc, Dijon, France.

ELIGIBILITY:
Inclusion Criteria:

* Women followed for breast cancer in Georges Francois Leclerc Center
* Neoadjuvant chemotherapy
* Age >= 18

Exclusion Criteria:

* Males
* Metastatic breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non metastatic breast cancer who received neoadjuvant chemotherapy prior to tumor surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-09-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 5 years
  Overall survival and evolution over years

SECONDARY OUTCOMES:
Collection of patient and treatment characteristics | 5 years
  Collection of patient and treatment characteristics over years, to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Locations (1):
- Methodology, Biostatistics and Data Management Unit, Dijon, France

IPD SHARING:
Plan to Share IPD: No